CLINICAL TRIAL: NCT00286130
Title: A Randomised, Open-label Phase II Study Evaluating the Efficacy and Safety of Folfox6 + Cetuximab as First-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy of Folfox6 + Cetuximab Versus Folfiri +Cetuximab in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/Core 1.2.001; EUDRACT number 2004-002391-42
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; FOLFOX 6; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX 6 (Active Comparator): FOLFOX 6:
  * Oxaliplatin 100 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks:
  Interventions: Drug: Cetuximab, Oxaliplatin, Leucovorin, 5FU, Irinotecan; Drug: FOLFOX 6
- FOLFIRI (Active Comparator): FOLFIRI:
  * Irinotecan 180 mg/m² day 1 concurrent with
  * Leucovorin 400 mg/m² followed by
  * Bolus 5FU 400 mg/m², followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  Interventions: Drug: Cetuximab, Oxaliplatin, Leucovorin, 5FU, Irinotecan; Drug: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab, Oxaliplatin, Leucovorin, 5FU, Irinotecan
Drug: FOLFOX 6 — FOLFOX 6:
  * Oxaliplatin 100 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks:
  Arms: FOLFOX 6
Drug: FOLFIRI — FOLFIRI:
  * Irinotecan 180 mg/m² day 1 concurrent with
  * Leucovorin 400 mg/m² followed by
  * Bolus 5FU 400 mg/m², followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  Arms: FOLFIRI

SUMMARY:
In Patients with metastatic colorectal cancer the following treatments first-line Folfiri+Cetuximab first-line Folfox6 + Cetuximab will be concerning efficacy and safety.

The trial compares Folfiri + Cetuximab and Folfox6 + Cetuximab concerning efficacy and safety as first

DETAILED DESCRIPTION:
The multicenter randomized phase II study will enroll a target of approximately 150 first-line patients with metastatic CRC.

EGFR expression is not required for study entry, however, the EGFR status will be measured retrospectively.

Patients are randomized to Arm A or Arm B. Arm A: FOLFOX 6 in combination with cetuximab Arm B: FOLFIRI in combination with cetuximab. Both efficacy and safety data will be collected. The investigators will assess response to treatment at 6 weeks, 12 weeks and thereafter every 12 weeks based on imaging Following permanent treatment cessation (stop of all study treatments) patients will be followed-up for.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* Metastatic colorectal carcinoma not suitable for curative-intent resection
* Availability of tumor sample (or able and willing to provide tumor sample) for EGFR assessment
* Presence of at least one lesion measurable unidimensional by CT scan or MRI (Target lesion(s) must not lie within an irradiated area)
* ECOG performance status of < 2 at study entry

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous chemotherapy for metastatic CRC or adjuvant therapy with oxaliplatin or irinotecan. Adjuvant therapy with 5 FU or derivatives is allowed if the chemotherapy treatment free interval is > 6 months
* Surgery (excluding diagnostic biopsy) or irritation within 4 weeks prior to study entry
* Cocurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to entry
* Previous exposure to EGFR-pathway targeting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
the percentage of patients surviving without disease progression in each arm at 9 months

SECONDARY OUTCOMES:
PFS rates at 3,6,12 months
Response rates
Overall survival (OS) in each arm
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Werner Scheithauer, MD, Principal Investigator — Dep. of Internal Medicine I, Medical University of Vienna
Locations (27):
- Austria (2):
  - LKH Leoben, Abt. für Innere Medizin, Leoben, Styria
  - Univ. Klinik für Innere Medizin I, Vienna
- Institute of Oncology, Sarajevo, Bosnia and Herzegovina
- Bulgaria (2):
  - University Hospital "Queen Joanna", Sofia
  - SBALO National Oncology Center, Sofia
- Croatia (2):
  - University Hospital for Tumors, Zagreb
  - University Hospital Rebro, Zagreb
- Bank of Cyprus Oncology Center, Nicosia, Cyprus
- Czechia (2):
  - Univ. Hospital Brno, Dept. Of Clinical Oncology, Brno
  - Charles University Prague, Dep. of Oncology, Prague
- Hungary (3):
  - National Medical Center, Budapest
  - Markusovsy Hospital, Szomathely
  - Csolnoky Ferenc County Hospital, Veszprém
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Souraski Medical Center, Tel Aviv
- Portugal (5):
  - Hospital Amadora Sintra, Servico de Oncologia, Amadora
  - Hospital de Beja, Beja
  - Hospital Distrital de Faro, Faro
  - Hospital Geral de Sto. António, Porto
  - Hospital San Teotóno -, Viseu
- Romania (2):
  - Institutul Oncologic Bucuresti, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
- National Cancer Institute, Bratislava, Slovakia
- Institute of Oncology, Ljubljana, Slovenia
- Turkey (Türkiye) (3):
  - Ankara Hacettepe University, Oncology Unit, Ankara
  - Gazi University Medical Faculty, Ankara
  - 9 Eyul University Medical Faculty, Dep of Oncology, Izmir